CLINICAL TRIAL: NCT00620347
Title: A Phase II Study of Sunitinib as a Second-line Treatment for Patients With Recurrent Small Cell Lung Cancer.
Brief Title: Sunitinib as a Second-line Treatment for Patients With Recurrent Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Center, Korea (Other Government)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Ji-youn Han, Head, Center for Lung Cancer, National Cancer Center, Korea
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCCTS-07-285
Record Dates: First submitted 2008-01-25; First posted 2008-02-21 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2013-06

CONDITIONS: Lung Cancer
Keywords: SCLC (small cell lung cancer); ED (extensive disease); RR (response rate)
MeSH Terms: conditions — Lung Neoplasms; Small Cell Lung Carcinoma | interventions — Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single arm (Experimental): Single arm (sunitinib arm) until PD, unacceptable toxicity, patients refused
  Interventions: Drug: sunitinib

INTERVENTIONS:
Drug: sunitinib — sunitinib (50mg/day, 4weeks on, 2 weeks off) Repeat every 6 weeks. Treatment will continue until disease progression, unacceptable toxicity, or patients' refusal.

SUMMARY:
the investigators will conduct a phase II trial to evaluate the efficacy and toxicity of Sunitinib in patients with recurrent SCLC.

DETAILED DESCRIPTION:
Chemotherapy is the primary treatment option for patients with small cell lung cancer, leading to a 5-year survival of about 20% in limited disease (LD), and less than 5% in extensive disease (ED). Although initial tumor response rate to chemotherapy is very high (up to 96% for LD and up to 65% in ED), SCLC relapses in approximately 4 months in ED and 12 months in LD adn despite the administration of second-line chemotherapy, the overall median survival of patients with limited and extensive disease is approximately 18 and 9 months, respectively. In the setting of second-line therapy, response rates to chemotherapy range between 15 and 25%, with median survival in the range of 4-6 months. Second-line therapeutic options include cyclophosphamide, doxorubicin and vincristine (CAV) given every 3 weeks or topotecan, which have similar response rates, time to progression and survival in the two treatment arms (topotecan 24%, 13 and 24.7 weeks; CAV 18%, 12 and 22 weeks, respectively). However, both treatments however have substantial toxicities, with 9% of patients on trial withdrawing for toxicity reasons. Treatment-associated mortality was as high as 4.7% (possibly and definitely related), and many patients required transfusion support. Thus, while these treatments have acceptable activity second-line, more active and less toxic treatments are required for this patient population.Tyrosine kinase inhibitors have become a promising new class of anti-cancer agents owing to the importance of their targets in tumor proliferation, survival (apoptosis), angiogenesis, motility, and metastasis Among the most important receptor tyrosine kinases that regulate tumor angiogenesis are the vascular endothelial growth factor receptor 2 (VEGFR2/Flk-1/KDR), PDGFR, and the fibroblast growth factor (FGF) receptor family. These receptors belong to the split-kinase domain superfamily, which also includes Kit, the receptor for stem cell factor (SCF). Kit is frequently expressed in multiple hematologic and non-hematologic malignancies. It can also be activated in an autocrine fashion by coexpression with SCF, as is the case in SCLC, where approximately 70% of tumors and cell lines coexpress Kit and SCF at some level. Inhibition of Kit using small molecule inhibitors results in growth inhibition of multiple SCLC cell lines. Sunitinib, a novel small molecule receptor tyrosine kinase inhibitor with direct antitumor as well as antiangiogenic activity via targeting the vascular endothelial growth factor (VEGF), platelet-derived growth factor (PDGF), KIT, and FLT3 receptor tyrosine kinases, which showed anti-tumor activity in mouse xenograft model of SCLC. Therefore, the investigators will conduct a phase II trial to evaluate the efficacy and toxicity of Sunitinib in patients with recurrent SCLC.-Single arm

-Sunitinib(50mg/day, 4weeks on, 2 weeks off) Repeat every 6 weeksTreatment will continue until disease progression, unacceptable toxicity, or patients' refusal

ELIGIBILITY:
Inclusion Criteria:

1. Histologic or cytologic confirmed SCLC
2. Clinically diagnosed ED-SCLC according to sixth Edition of the AJCC cancer staging manual
3. Progression during or after prior first line chemotherapy.
4. Resolution of all acute toxic effects of prior therapy or surgical procedure to grade ≤ 1 (except alopecia)
5. Prior radiation therapy excluded lung is allowed.
6. No other forms of cancer therapy, such as chemotherapy, radiation, immunotherapy for at least 3 weeks before the enrollment in study.
7. Performance status of 0, 1, 2 on the ECOG criteria.
8. Tumor work-up: within 4weeks prior 1st day of treatment: chest X-ray; CT of chest, liver, and adrenal glands; bone scan; brain MRI
9. At least one uni-dimensionally measurable lesion meeting Response Evaluation Criteria in Solid Tumors.
10. Estimated life expectancy of at least 12 weeks.
11. Patient compliance that allows adequate follow-up.
12. Adequate organ function for chemotherapy
13. Adequate cardiac function: normal EF by Echocardiography
14. No ischemic heart disease or cardiac dysrhythmia.
15. Normal QTc interval
16. Normal thyroid function.
17. Informed consent from patient or patient's relative.
18. Males or females at least 18 years of age.
19. If female: childbearing potential either terminated by surgery, radiation, or menopause, or attenuated by use of an approved contraceptive method (intrauterine device [IUD], birth control pills, or barrier device) during and for 3 months after trial. If male, use of an approved contraceptive method during the study and 3 months afterwards. Females with childbearing potential must have a urine negative HCG test within 7 days prior to the study enrollment.

Exclusion Criteria:

1. Diagnosis of any second malignancy within the past 3 years, except basal cell carcinoma, squamous cell skin cancer, or in situ carcinoma that has been adequately treated with no evidence or recurrent disease for 12 months
2. NCI CTCAE grade ≥ 2 neuropathy from any cause
3. Ongoing treatment with therapeutic doses of coumarin derivatives, such as warfarin, (low dose Coumadin® up to 2 mg PO daily for deep vein thrombosis prophylaxis is allowed)
4. Uncontrolled brain metastases, spinal cord compression, carcinomatous meningitis, or leptomeningeal disease. Patients should have completed surgery or radiation therapy for existing brain metastases, should not have documented increase in size over the previous 3 months and should be asymptomatic off steroids
5. Any of the following within the 12 months prior to starting study treatment: myocardial infarction, sever/unstable angina, coronary/peripheral artery bypass graft, congestive heart failure, cerebrovascular accident including transient ischemic attack, or pulmonary embolus
6. NCI CTCAE Grade 3 hemorrhage < 4 weeks of starting study treatment
7. Hypertension (>150/100 mg Hg) that cannot be controlled with standard antihypertensive agents
8. Ongoing cardiac dysrhythmias of grade ≥ 2, atrial fibrillation of any grade, or QTc interval > 450 msec for males or > 470 msec for female
9. Known human immunodeficiency virus (HIV) seropositivity
10. Pregnancy or breastfeeding. All female patients with reproductive potential must have a negative pregnancy test (serum or urine) within 7 days prior to enrolment
11. Other severe acute or chronic medical or psychiatric condition, or laboratory abnormality that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results, and in the judgment of the investigator would make the patient inappropriate for entry into this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2008-03; Primary Completion 2012-02 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Tumor response rate | at 4week and every 8 weeks
  The response rate will be determined by the number of patients with complete and partial responses according to RECIST criteria.

SECONDARY OUTCOMES:
Overall survival | every 8 weeks
  Survival time will be calculated from the date of study treatment start to the date of death (or date last seen).
Progression-Free Survival | at 4 week and every 8 weeks
  Progression free survival will be calculated from the date of study treatment start to the first objective documentation of progressive disease or death.
Toxicity | every 4 weeks
  Safety will be evaluated by the frequency, severity, and relationship of adverse events graded by NCI Common Toxicity Criteria (CTC) version 3.0 that occur during the treatment and follow-up periods.

CONTACTS AND LOCATIONS:
Overall Officials: Ji-Youn Han, M.D.,Ph.D., Principal Investigator — National Cancer Center, Korea
Locations (1):
- National Cancer Center, Korea, Goyang-si, Gyeonggi-do, South Korea

REFERENCES:
- [Derived] Han JY, Kim HY, Lim KY, Han JH, Lee YJ, Kwak MH, Kim HJ, Yun T, Kim HT, Lee JS. A phase II study of sunitinib in patients with relapsed or refractory small cell lung cancer. Lung Cancer. 2013 Feb;79(2):137-42. doi: 10.1016/j.lungcan.2012.09.019. Epub 2012 Nov 20. PMID 23182663